CLINICAL TRIAL: NCT06640088
Title: Determining ICU Staffs Conceptions, Opinions, Views, Experiences and Reflection of Brain Death and Organ Donation
Acronym: DISCOVER
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2024-01116, am24Sutter
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Brain Death
Keywords: Organ Donation; Intensive Care Unit
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to gather information regarding the individual perceptions, opinions, beliefs, and conceptual understanding of healthcare professionals working in the intensive care units at the University Hospital Basel and to determine associations of individual beliefs, personal, educational, and professional experiences with individual perceptions, opinions, and conceptual understanding regarding brain death and organ donation.

DETAILED DESCRIPTION:
To achieve the study objectives, the investigator will employ a questionnaire-based survey administered to the consenting/participating nurses and physicians. The questionnaire will address various aspects related to personal background, religious affiliation, beliefs about life after death, the conceptual understanding of brain death and organ donation, as well as experiences and opinions related to these topics.

ELIGIBILITY:
Inclusion Criteria:

* Consenting nurses and physicians currently working in the intensive care unit (ICU) at the University Hospital Basel
* Only nurses and physicians consenting to participate will be included

Exclusion Criteria:

* Nurses and physicians not currently working (any more) in the intensive care unit (ICU) at the University Hospital Basel
* Nurses and physicians who do not consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible healthcare professionals in the ICU at the University Hospital Basel
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Information on individual perceptions regarding brain death and organ donation | at baseline
  Descriptive analyses will be performed to identify individual perceptions
Information on individual opinions regarding brain death and organ donation | at baseline
  Descriptive analyses will be performed to identify individual opinions
Information on individual beliefs regarding brain death and organ donation | at baseline
  Descriptive analyses will be performed to identify individual beliefs
Information on conceptual understanding regarding brain death and organ donation | at baseline
  Descriptive analyses will be performed to identify conceptual understanding
Identification of interprofessional variations | at baseline
  Descriptive analyses will be performed to identify interprofessional variations

CONTACTS AND LOCATIONS:
Overall Officials: Raoul C. Sutter, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland